CLINICAL TRIAL: NCT05599867
Title: Biological Therapy in Patients With Inflammatory Bowel Disease :Laboratory ,Endoscopic and Quality of Life Assessment
Brief Title: Biological Therapy in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: Amany123
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Quality of Life
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: quality of life — to assess quality among patients with patients with IBD

SUMMARY:
Inflammatory bowel disease (IBD) is characterised by chronic, relapsing inflammation of the intestinal mucosa and an inability to down regulate the inflammatory immune response once activated. IBD encompasses ulcerative colitis (UC), Crohn's disease (CD) and indeterminate colitis which is not clearly diagnosed as UC or CD. The peak age of onset of IBD is 15 to 30 years, with a second smaller peak occurring between 50 and 70 years of age

DETAILED DESCRIPTION:
The incidence of IBD is rapidly increasing in newly industrialized countries strongly implicating environmental factors. The pathogenesis of IBD is not fully understood, but key influences are thought to include genetics, environmental factors, immune response, and gut microbiota.It is recognised that the availability of vitamin D is important in regulating gut mucosal immunity; with studies suggesting that vitamin D may affect gut epithelial integrity, innate immune barrier function, and the development and function of T cells The predominant symptoms of IBD are diarrhea, abdominal pain, gastrointestinal bleeding, weight loss, malnutrition and fatigue which can substantially impact a patient's quality of life (QoL), largely due to the psychosocial impact of symptoms. A survey of IBD outpatients found that concerns about loss of bowel control, producing unpleasant odours, achieving their full potential in the workplace, feeling dirty or smelly, and issues with sexual relationships, ranked highly for both UC and CD

ELIGIBILITY:
Inclusion Criteria:

- Any patient who is above age of 18 years old and diagnosed to have IBD (UC and/or CD) and eligible for biological therapy will be recruited in the study.

Exclusion Criteria:

* Patients with IBD who aren't eligible to biological therapy
* Pregnant patients with IBD
* Patients with IBD who are under age of 18 years old
* Patient's refusal

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Diagnosis of IBD will be based on combination between clinical, laboratory, radiological, endoscopic and/or histopathological data Indications of biological therapy are based on the current diagnostic and treatment recommendations of Epidemiological Committee of European Crohn's and Colitis Organization (ECCO). In most countries, moderate to severe luminal CD, or perianal or fistulising CD, or moderate to severe UC patients with immunosuppressant or corticosteroid refractory disease, or those with intolerance or contraindication to conventional therapies are eligible to be treated with biological therapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
quality of life in patients with IBD after biological therapy | one year
  we use The SF-36 form

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abu-Elfatth, Principal Investigator — Assiut University
Locations (1):
- Ahmed, Al Minyā, Alminya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
with special request

REFERENCES:
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646